CLINICAL TRIAL: NCT04763746
Title: The Measurement of VItal SIgns by Lifelight® Software in comparisON to the Standard of - Multi-site Development: The VISION-MD Study
Brief Title: The Measurement of VItal SIgns by Lifelight® Software in comparisON to the Standard of Care - Multi-site Development
Acronym: VISION-MD
Status: Completed | Type: Observational
Sponsor: Xim Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: IRAS: 289242
Record Dates: First submitted 2021-02-08; First posted 2021-02-21 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2023-01

CONDITIONS: Respiratory Disorder; Diabetes; Cardiovascular Diseases; Critical Care; Trauma and Emergency Care; Primary Care
Keywords: vital signs; innovation; lifelight; blood pressure; oxygen saturation; contactless; rPPG
MeSH Terms: conditions — Respiration Disorders; Diabetes Mellitus; Cardiovascular Diseases; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Sub-protocol 1: Blood pressure, oxygen saturation and heart rate measured from participants selected because of their blood pressure.
  Within each study session, participants will have their blood pressure, oxygen saturation and heart rate measured three times using standard-of-care equipment and methods. At the same time, video of the participant's face will be captured using the Data Collect app running on a tablet positioned opposite them.
  Interventions: Device: Lifelight Data Collect Sub-protocol 1
- Sub-protocol 2: Respiratory rate and oxygen saturation measured from any participant.
  Within each study session, participants will have their respiratory rate and oxygen saturation measured twice using standard-of-care equipment and methods. At the same time, video of the participant's face will be captured using the Data Collect app running on a tablet positioned opposite them.
  Interventions: Device: Lifelight Data Collect Sub-protocol 2
- Sub-protocol 3: Oxygen saturation measured from participants expected to have low oxygen saturation.
  Within each study session, participants will have their oxygen saturation measured twice using standard-of-care equipment. At the same time, video of the participant's face will be captured using the Data Collect app running on a tablet positioned opposite them.
  Interventions: Device: Lifelight Data Collect Sub-protocol 3
- Sub-protocol 4: Blood pressure, heart rate, respiratory rate and oxygen saturation measured from adults lacking capacity.
  Within each study session, participants will have their blood pressure, heart rate, respiratory rate and oxygen saturation measured three times using standard-of-care equipment and methods. At the same time, video of the participant's face will be captured using the Data Collect app running on a tablet positioned opposite them.
  Interventions: Device: Lifelight Data Collect Sub-protocol 4

INTERVENTIONS:
Device: Lifelight Data Collect Sub-protocol 1 — Study nurse 1 will announce when the 60-second period of Lifelight® measurement begins and ends, guided by the timer on the software. They will observe the oxygen saturation measurements during this 60-second measurement period, noting down the first reading displayed at 0, 30 and 60 seconds. The three oxygen saturation readings should be averaged to generate a single, average oxygen saturation reading.
  Study nurse 2 will operate the automatic sphygmomanometer upon hearing from study nurse 1 that the 60-second measurement period has begun. Study nurse 2 will then spend the remaining measurement period observing the heart rate measurements and note the reading displayed after 0, 30 and 60 seconds. The three heart rate readings should be averaged to generate a single, average heart rate reading.
  This sub-protocol will be repeated twice more to generate three sets of blood pressure, heart rate and oxygen saturation measurements and three concurrent video datasets.
  Groups: Sub-protocol 1
Device: Lifelight Data Collect Sub-protocol 2 — Study nurse 1 will announce when the 60-second period of Lifelight® measurement begins and ends, guided by the timer on the software. They will observe the oxygen saturation measurements during this 60-second measurement period noting down the first reading displayed at 0, 30 and 60 seconds timepoints. The three oxygen saturation readings should be averaged to generate a single, average oxygen saturation reading.
  Study nurse 2 will be directed by the announcement of study nurse 1 to begin and end manually counting observed inspirations by watching chest rises throughout the full 60-second period. According to the results of the quality improvement initiative, Study nurse 2 may place their hand on the participant's chest to increase the accuracy of their manual counting.
  This sub-protocol will be repeated once more to generate two sets of respiratory rate and oxygen saturation measurements and two concurrent video datasets.
  Groups: Sub-protocol 2
Device: Lifelight Data Collect Sub-protocol 3 — The study nurse will observe the oxygen saturation measurements during this 60-second measurement period indicated by the timer on the software. They will note down the first reading displayed after 0, 30 and 60 seconds. The three oxygen saturation readings should be averaged to generate a single, average oxygen saturation reading for the 60-second period.
  This sub-protocol will be repeated once more to generate two sets of oxygen saturation measurements and two concurrent video datasets.
  Groups: Sub-protocol 3
Device: Lifelight Data Collect Sub-protocol 4 — Study nurse 1 will announce when the 60-second period of Lifelight® measurement begins and ends, guided by the timer on the software. They will manually count observed inspirations by watching chest rises throughout the 60-second period. They may place their hand on the participant's chest to increase the accuracy of manual counting.
  Study nurse 2 will operate a standard automatic sphygmomanometer and clinical finger clip sensor upon hearing from Study nurse 1 that the 60-second measurement period has begun. Study nurse 2 will then spend the remaining measurement period observing these measurements and note the readings displayed after 0, 30 and 60 seconds. The three heart rate and three oxygen saturation readings will each be averaged to generate a single, average reading.
  This sub-protocol will be repeated twice more to generate three sets of blood pressure, heart rate, respiratory and oxygen saturation measurements and three concurrent video datasets.
  Groups: Sub-protocol 4

SUMMARY:
AIM: To advance the development and accuracy of the Lifelight® app for the measurement of vital signs, therefore developing a non-invasive and easy-to-perform means of measuring vital signs which can be implemented across a wide range of settings, both within hospitals and out in the community.

METHOD: Lifelight® is a computer program ("app") for measuring vital signs which can be used on smart devices that contain a camera. It is able to measure all of the vital signs by measuring very small changes in skin colour that occur each time the heart beats. This means that it does not need to touch the patient. The investigators believe this could be an effective way of measuring vital signs, especially during the COVID-19 pandemic when prevention of cross-contamination between patients is essential. Patients are also likely to be reassured by a contactless approach. The app uses data from looking at a person's face to calculate the vital signs. This is possible because there are tiny changes in facial skin that occur each time the heart beats.

The investigators believe Lifelight® could be an effective way of measuring vital signs. The app is still under development, which means that it is still "learning" the best match between the information it collects from the face and the values of vital signs measured using the standard equipment. The app should become more accurate in calculating the vital signs as it sees more and more information from patients.

So far, the app has seen data from inpatients, outpatients, patients attending GP surgeries and healthy people. This has improved its accuracy in measuring vital signs. However, the app needs to see more information so that it can be sufficiently accurate for specific clinical applications such as long-term monitoring of hypertension. To do this, it particularly needs to see information from people with abnormal blood pressures and blood oxygen levels. In order to capture the full range of observations, the app will need to be trialled with some of the most critically ill patients - some of these will not have capacity to consent to participation in the study. It also needs to see more data from people with different skin tones so the investigators can be sure it is accurate for all patients.

To do this, the investigators will recruit people who are attending one of two hospitals, either as an inpatient, an outpatient, a friend/relative of a patient, or a member of hospital staff. The exact number will depend on how quickly the app "learns" and how many of the vital signs are outside of the normal range. The investigators will take the participant's vital signs using standard clinical equipment whilst recording a video of their face. The investigators will use most of these measurements and video to teach the app how to become more accurate at measuring vital signs. The investigators will keep the remaining data separate and use it to test how accurate the app is. All of the data will be kept securely.

The investigators will also collect feedback from participants and healthcare staff on their experiences using the app and information that allows us to assess whether there are any savings to the healthcare economy through use of this technology.

DETAILED DESCRIPTION:
Following informed consent, the study staff member will complete a very brief set of demographic and medical history questions, limited to the presence or absence of medical problems and treatment for them.

Participants with capacity to consent will be recruited into either Sub-protocol 1, 2 or 3 on the basis of which vital signs are expected to be abnormal. Participants who lack capacity to consent to take part in the study will be recruited into Sub-protocol 4.

* Sub-protocol 1 participants will have blood pressure, oxygen saturation and heart rate measured.
* Sub-protocol 2 participants will have respiratory rate and oxygen saturation measured.
* Sub-protocol 3 participants will have oxygen saturation measured.
* Sub-protocol 4 participants will have blood pressure, heart rate, respiratory rate and oxygen saturation measured.

Participants may also be recruited to a sub-protocol on the basis of their skin tone. This is because there are targets within Sub-protocols 1, 2 and 3 related to skin tone.

Not all vital signs are collected in all participants to focus study nurse attention on fewer tasks and to avoid collection of data that is not subsequently used to meet the study objectives. This approach should help to keep all aspects of data collection as high quality as possible and is consistent with the GDPR requirement of data minimisation.

For all Sub-protocol 1, 2, 3 and 4 participants, the study team will complete a set of pre-measurement observation questions. Background luminosity will be measured using a handheld lux meter. The staff member will then prepare for and take the participant's routine observations using standard clinical equipment during the same 60-second period that video is captured of the participant's face using the Data Collect app. Best efforts will be made to adhere to the Lifelight® measurement conditions listed in Appendix B. These measurements and video capture will be repeated once more in the case of Sub-protocols 2 and 3, and twice more in the case of Sub-protocols 1 and 4. Once measurements are concluded, the study staff member will complete the post-measurement observation questions. In all cases, the cleaning protocol outlined in Appendix D will be adhered to after each study session.

A selection of Sub-protocol 1, 2 and 3 participants will be asked to complete a questionnaire related to vital sign monitoring and their preference of Lifelight® or other technologies for measuring vital signs.

ELIGIBILITY:
Inclusion Criteria:

* 16 years old or above

Exclusion Criteria:

* None

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Inpatients, outpatients, staff and healthy participants - adults only (16+)
Sampling Method: Non-Probability Sample
Enrollment: 1869 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Train Lifelight algorithms across more extensive clinical ranges, including patients with an blood oxygen saturation of <92%, to reach closer to a performance target of 4% maximum error tolerance. | 12 months
Train Lifelight algorithms across more extensive clinical ranges, including patients with a systolic blood pressure of <90 or >180 mmHg, to progress towards British Hypertension Society Grade C and a standard deviation performance target of <8mmHg. | 12 months
Train Lifelight algorithms across more extensive clinical ranges, including patients with a diastolic blood pressure of >110 mmHg, to improve Lifelight's British Hypertension Society Grade B grading and standard deviation performance target of <8mmHg | 12 months
Train Lifelight algorithms across more extensive clinical ranges, including patients with a pulse of <40bpm or >120bpm, to reach closer to the indicative performance target of an RMSE of 3bpm or less. | 12 months
Train Lifelight algorithms across more extensive clinical ranges, including patients with a respiration rate of >25 rpm, to reach closer to the indicative performance target of a 5 breath per minute maximum error tolerance. | 12 months
Train Lifelight algorithms on a more diverse population, including patients with Fitzpatrick scale 1, 4, 5 and 6 skin tones. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Laura Wiffen, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (1):
- Portsmouth Hospitals NHS Trust, Portsmouth, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kiddle A, Barham H, Wegerif S, Petronzio C. Dynamic Region of Interest Selection in Remote Photoplethysmography: Proof-of-Concept Study. JMIR Form Res. 2023 Mar 30;7:e44575. doi: 10.2196/44575. PMID 36995742
- [Derived] Wiffen L, Brown T, Brogaard Maczka A, Kapoor M, Pearce L, Chauhan M, Chauhan AJ, Saxena M; Lifelight Trials Group. Measurement of Vital Signs by Lifelight Software in Comparison to Standard of Care Multisite Development (VISION-MD): Protocol for an Observational Study. JMIR Res Protoc. 2023 Jan 11;12:e41533. doi: 10.2196/41533. PMID 36630158